CLINICAL TRIAL: NCT05801705
Title: Comparative Evaluation of Efficacy and Safety of Toremifene, Tamoxifen, and Aromatase Inhibitor Plus Ovarian Suppression in Hormone Receptor-Positive Early Breast Cancer Among Non-Low-Risk Premenopausal Women: A Real-World Study
Brief Title: Comparative Evaluation of Efficacy and Safety of Toremifene, Tamoxifen, and Aromatase Inhibitor Plus Ovarian Function Suppression in Hormone Receptor-Positive Early Breast Cancer Among Non-Low-Risk Premenopausal Women: A Real-World Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Gong, professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2022-445-02
Record Dates: First submitted 2023-03-26; First posted 2023-04-06 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Hormone-receptor-positive Breast Cancer; Premenopausal Breast Cancer; Breast Cancer Patients at Intermediate to High Risk; Ovarian Function Suppression Combined With Aromatase Inhibitor or Tamoxifen or Torimefen
MeSH Terms: interventions — Aromatase Inhibitors; Ovariectomy; Gonadotropin-Releasing Hormone; Tamoxifen; Toremifene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OFS+AI: patients undergoing ovarian function suppression (OFS) combined with aromatase inhibitor (AI)
  Interventions: Drug: Aromatase inhibitor; Procedure: ovarian function suppression (Oophorectomy, Ovarian irradiation, Gonadotropin-releasing hormone agonist)
- OFS+TAM: patients undergoing ovarian function suppression (OFS) combined with tamoxifen (TAM)
  Interventions: Procedure: ovarian function suppression (Oophorectomy, Ovarian irradiation, Gonadotropin-releasing hormone agonist); Drug: Tamoxifen
- OFS+TOR: patients undergoing ovarian function suppression (OFS) combined with torimifene (TOR)
  Interventions: Procedure: ovarian function suppression (Oophorectomy, Ovarian irradiation, Gonadotropin-releasing hormone agonist); Drug: toremifene

INTERVENTIONS:
Drug: Aromatase inhibitor — Aromatase inhibitor includes Arimidex, Aromasin, Femara.
  Groups: OFS+AI
Procedure: ovarian function suppression (Oophorectomy, Ovarian irradiation, Gonadotropin-releasing hormone agonist) — Gonadotropin-releasing hormone agonist includes Buserelin, Goserelin, Leuprorelin, Nafarelin, Triptorelin
Drug: Tamoxifen — tamoxifen,10mg, bid
  Groups: OFS+TAM
Drug: toremifene — toremifene, 60 mg, qd
  Groups: OFS+TOR

SUMMARY:
This study aims to enroll premenopausal patients, with early breast cancer who are non-low-risk and hormone receptor-positive and have undergone prior surgical intervention at the Breast Cancer Center of Sun Yat-sen Memorial Hospital, Sun Yat-sen University. These participants, receiving tamoxifen (TAM), toremifene (TOR), or aromatase inhibitors (AI) as adjuvant endocrine therapy and undergoing ovarian function suppression (OFS) treatment, will be divided into three groups, namely TOR+OFS, TAM+OFS, AI+OFS. The study will compare the efficacy and safety of TOR+OFS to that of TAM+OFS or AI+OFS in premenopausal estrogen receptor-positive breast cancer patients by comparing the 5-year disease-free survival (DFS) and quality of life etc. The objective is to evaluate whether TOR+OFS is non-inferior to TAM+OFS or AI+OFS in this specific patient population.

DETAILED DESCRIPTION:
Selective estrogen receptor modulators (SERM), tamoxifen (TAM) and toremifene (TOR), have been proven to be effective in premenopausal estrogen receptor positive breast cancer patients with similar outcomes. In addition, many large-scale long-term follow-up clinical tials, such as ABCSG XII, SOFT, TEXT, ASTRRA, and ZIPP, have confirmed that premenopausal patients with hormone-receptor-positive breast cancer at intermediate to high risk could benefit from ovarian function suppression (OFS) combined with aromatase inhibitor (AI) or TAM. The Asian Breast Cancer Cooperative Group (ABCCG) also recommends OFS+TAM or OFS+AI for the treatment in this specific patient population. Notably, the therapeutic efficacy and safety profile of OFS in conjunction with TOR have yet to be investigated, nor has its comparative effectiveness with OFS plus TAM or OFS plus AI been established.

This study aims to enroll premenopausal patients, with early breast cancer who are non-low-risk and hormone receptor-positive and have undergone prior surgical intervention at the Breast Cancer Center of Sun Yat-sen Memorial Hospital, Sun Yat-sen University. These participants, receiving tamoxifen (TAM), toremifene (TOR), or aromatase inhibitors (AI) as adjuvant endocrine therapy and undergoing ovarian function suppression (OFS) treatment, will be divided into three groups, namely TOR+OFS, TAM+OFS, AI+OFS. The study will compare the efficacy and safety of TOR+OFS to that of TAM+OFS or AI+OFS in premenopausal estrogen receptor-positive breast cancer patients by comparing the 5-year disease-free survival (DFS) and quality of life etc. The objective is to evaluate whether TOR+OFS is non-inferior to TAM+OFS or AI+OFS in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged 18-60
2. Premenopausal patients with early hormone receptor-positive breast cancer at intermediate to high risk (Low risk is defined as having the following 6 items at the same time: lesion size (pT) in the specimen <= 2cm; histological grade 1; no vessel carcinoma embolus; ER and/or PR positive; HER2 gene without overexpression or amplification; age >=35 years old)
3. Completed radical surgery for breast cancer
4. Undergoing postoperative endocrine therapy (toremifene, tamoxifen, aromatase inhibitorI) at least five years at Sun Yat-sen Memorial Hospital of Sun Yat-sen University since 2010
5. Undergoing ovarian function suppression (Oophorectomy, Ovarian irradiation, Gonadotropin-releasing hormone agonist)

Exclusion Criteria:

1. Imaging or pathology suggestive of metastatic breast cancer (chest wall, lung, bone, liver, brain)
2. Patients with a second primary tumor
3. Hepatic insufficiency at baseline
4. Known history of psychotropic substance abuse or drug abuse;

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. Female, age ≥ 18
  2. Premenopausal patients with early hormone receptor-positive breast cancer at intermediate to high risk (Low risk is defined as having the following 6 items at the same time: lesion size (pT) in the specimen <= 2cm; histological grade 1; no vessel carcinoma embolus; ER and/or PR positive; HER2 gene without overexpression or amplification; age >=35 years old)
  3. Completed radical surgery for breast cancer
  4. Undergoing postoperative endocrine therapy (toremifene, tamoxifen, aromatase inhibitorI) at least five years at Sun Yat-sen Memorial Hospital of Sun Yat-sen University since 2010
  5. Undergoing ovarian function suppression (Oophorectomy, Ovarian irradiation, Gonadotropin-releasing hormone agonist)
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years
  The time from the beginning of treatment to the recurrence of the disease or death from any cause or the end of the visit
The score of life quality questionnaire assessed by SPF 36 | 1 month
  The score of SPF 36
The score of life quality questionnaire assessed by EQ-5D-5L | 1 month
  The score of EQ-5D-5L

SECONDARY OUTCOMES:
The incidence of adverse events | 5 years
  Incidence of adverse outcome events (such as musculoskeletal symptoms，osteoporosis, fragile, bone mineral density loss, hepatic insufficiency, dyslipidemia, endometrial hyperplasia, uterine fibroids, ovarian cyst, adenomyosis, hot flashes, night sweats etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Gong, docto, Study Chair — Sun Yat-sen Memorial Hospital of Sun Yat-sen Univeristy
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China